CLINICAL TRIAL: NCT03977519
Title: Effect of Manual Acupuncture Versus Transcutaneous Electric Nerve Stimulation for Primary Dysmenorrhea: a Randomized Controlled Trial
Brief Title: Effect of MA Versus TENS for Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Jingxue Yuan, Postgraduate of acupuncture department, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-176-KY
Record Dates: First submitted 2019-05-27; First posted 2019-06-06 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-06

CONDITIONS: Primary Dysmenorrhea
Keywords: primary dysmenorrhea; manual acupuncture; transcutaneous electric nerve stimulation; randomized controlled trial
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MA group (Experimental): Huatuo Brand needles (0.30×25mm,0.30×40mm or 0.30×75mm) will be used at EX-B8,BL32,SP8,and SP6.
  Interventions: Procedure: MA
- TENS group (Active Comparator): Huatuo Brand electrode patch (50mm×50mm) and the SDZ-V EA apparatus (Suzhou Medical Appliance) will be used to stimulate the area along the lower borders of the ribs and the upper borders of the hip crests on both sides.The parameters of the electric acupuncture apparatus：Continuous wave,the frequency is 100Hz, the current intensity is 2.5mA-5mA.
  Interventions: Procedure: TENS

INTERVENTIONS:
Procedure: MA — Huatuo Brand needles (0.30×25mm,0.30×40mm or 0.30×75mm) will be used.Participants will receive manual acupuncture for 30 minutes each time.After acupuncture,we will twist the needles every 10 minutes for about 30 seconds.The patients will be treated in their first day of dysmenorrhea, once a day for three consecutive days. And the treatments will last for three consecutive menstrual cycles.
  Arms: MA group
Procedure: TENS — Huatuo Brand electrode patch (50mm×50mm) and the SDZ-V EA apparatus (Suzhou Medical Appliance) will be used.Participants will receive transcutaneous electric nerve stimulation for 30 minutes each time.They will be treated in their first day of dysmenorrhea, once a day for three consecutive days. And the treatments will last for three consecutive menstrual cycles.
  Arms: TENS group

SUMMARY:
The trial aims to evaluate the effect of manual acupuncture versus transcutaneous electric nerve stimulation in treating primary dysmenorrhea.

DETAILED DESCRIPTION:
According to systematic reviews,manual acupuncture(MA) and high frequency transcutaneous electric nerve stimulation(TENS) had certain therapeutic effects on primary dysmenorrhea respectively.

In this trial, 84 patients with primary dysmenorrhea will be recruited and randomly allocated into MA group and TENS group. Patients in MA group will receive treatment at acupoints of Shiqizhui(EX-B8), Ciliao(BL 32),Diji(SP 8) and Sanyinjiao(SP 6) and those in TENS group will receive treatment at the area along the lower borders of the ribs and the upper borders of the hip crests on both sides. All patients, both in EA group and TENS group, will be treated in their first day of dysmenorrhea, once a day for three consecutive days. And the treatments will last for three consecutive menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Female;
2. Aged of 18 to 40 years;
3. Conforming to the criteria for the diagnosis of primary dysmenorrhea in the guideline developed by Society of Obstetricians and Gynaecologists of Canada（SOGC）in 2017.
4. With normal menstrual cycle(28±7 days) and normal menstrual period（3-7days）；
5. Menstrual mean pain score ≥4 on the numerical rating scale (NRS)；
6. To sign the informed consent and participate in the study voluntarily.

Exclusion Criteria:

1. Secondary dysmenorrhea;
2. Pregnant patients,lactating patients or patients preparing pregnancy.
3. Subjects with serious heart, liver, kidney damage or cognitive impairment, aphasia, mental disorders, or the inability to cooperate with the examination and treatment;
4. Subjects with coagulation dysfunction or anticoagulants such as warfarin and heparin have been used all the time;
5. Subjects installed with the cardiac pacemaker;
6. Those who have received relevant acupuncture, transcutaneous electric nerve stimulation and other treatment (except pain medication) the last three months;
7. Patients who may be allergic to electrodes.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with at least 50% reduction in mean pain intensity from baseline. | Baseline；At the end of menstrual period of Cycle 3(each menstrual period is about 3-7 days,each cycle is about 28 days)
  The pain intensity was measured by the Numerical Rating Scale (NRS), which is a valid measure of pain intensity with scores from 0 (no pain) to 10 (worst possible pain).Participants will be asked to rate their mean pain intensity on the days with pain during the third menstruation by selecting a single number from 0 to 10.The primary outcome is the proportion of patients with at least 50% reduction in mean pain intensity from baseline.

SECONDARY OUTCOMES:
Change of mean pain intensity from baseline measured by NRS. | Baseline；At the end of menstrual period of Cycle 1,Cycle 2,Cycle 3 and Cycle 6(each menstrual period is about 3-7 days,each cycle is about 28 days)
  The Numerical Rating Scale (NRS) is a valid measure of pain intensity with scores from 0 (no pain) to 10 (worst possible pain).Participants will be asked to rate their mean pain intensity on the days with pain during the menstruation by selecting a single number from 0 to 10.The outcome is the changed number of numerical rating scale(NRS)of mean pain intensity on the days with pain during the menstruation compared with baseline.
Change of the most severe pain intensity measured by NRS. | Baseline；At the end of menstrual period of Cycle 1,Cycle 2,Cycle 3 and Cycle 6(each menstrual period is about 3-7 days,each cycle is about 28 days)
  The Numerical Rating Scale (NRS) is a valid measure of pain intensity with scores from 0 (no pain) to 10 (worst possible pain).Participants will be asked to rate their worst pain intensity during the menstruation by selecting a single number from 0 to 10.The outcome is the changed number of numerical rating scale(NRS)of worst pain intensity during the menstruation compared with baseline.
Change of Cox Menstrual Symptom Scale(CMSS) | Baseline；At the end of menstrual period of Cycle 1,Cycle 2,Cycle 3 and Cycle 6(each menstrual period is about 3-7 days,each cycle is about 28 days)
  CMSS is a tool for evaluating patients' symptom integrally which consists of 17 items or symptoms.In severity evaluation,each symptom is scored in five levels: 0 represent symptoms not noticeable;1, slightly bothersome;2, moderate bothersome; 3, severely bothersome;4, very severely bothersome.
  In the duration of the evaluation,each variable is scored in five grades by the retained time of symptom: 0 score denote did not occur;1, lasted less than 3h; 2, lasted 3 to 7h;3, lasted an entire day;and 4, lasted several days.
Change of sick leave from baseline | Baseline；At the end of menstrual period of Cycle 1,Cycle 2,Cycle 3 and Cycle 6(each menstrual period is about 3-7 days,each cycle is about 28 days)
  Sick leave(the days of absence from work or school due to menstrual pain) will be recorded by participates.
Change of pain duration from baseline | Baseline；At the end of menstrual period of Cycle 1,Cycle 2,Cycle 3 and Cycle 6(each menstrual period is about 3-7 days,each cycle is about 28 days)
  Participates will be asked to record the pain duration(number of days with pain) in the menstrual period.

OTHER OUTCOMES:
Pain medication intake | At the end of menstrual period of Cycle 1,Cycle 2,Cycle 3 and Cycle 6(each menstrual period is about 3-7 days,each cycle is about 28 days)
  Participates will be asked to record the doses and frequency of pain-relief drugs they have taken.
Patients' satisfaction towards treatment. | At the end of menstrual period of Cycle 3 and Cycle 6(each menstrual period is about 3-7 days,each cycle is about 28 days)
  Patients will be asked to choice the satisfaction towards treatment.The satisfaction consist of dissatisfaction,a little satisfaction,moderate satisfaction,greater satisfaction and very satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jingxue Yuan, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burnett M, Lemyre M. No. 345-Primary Dysmenorrhea Consensus Guideline. J Obstet Gynaecol Can. 2017 Jul;39(7):585-595. doi: 10.1016/j.jogc.2016.12.023. PMID 28625286
- [Background] Blodt S, Pach D, Eisenhart-Rothe SV, Lotz F, Roll S, Icke K, Witt CM. Effectiveness of app-based self-acupressure for women with menstrual pain compared to usual care: a randomized pragmatic trial. Am J Obstet Gynecol. 2018 Feb;218(2):227.e1-227.e9. doi: 10.1016/j.ajog.2017.11.570. Epub 2017 Nov 15. PMID 29155036
- [Background] Woo HL, Ji HR, Pak YK, Lee H, Heo SJ, Lee JM, Park KS. The efficacy and safety of acupuncture in women with primary dysmenorrhea: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Jun;97(23):e11007. doi: 10.1097/MD.0000000000011007. PMID 29879061
- [Background] Proctor ML, Smith CA, Farquhar CM, Stones RW. Transcutaneous electrical nerve stimulation and acupuncture for primary dysmenorrhoea. Cochrane Database Syst Rev. 2002;2002(1):CD002123. doi: 10.1002/14651858.CD002123. PMID 11869624